CLINICAL TRIAL: NCT04356209
Title: Improving Theempowerment in Patients With Severe Breast Fibrosis Radio-induced Treated by Pravastatin : Benefit of e-PROs (Electronic " Patient Reported Outcome ") on Breast-related Quality of Life
Acronym: PRAVACUR-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2019-02 PRA
Record Dates: First submitted 2020-04-14; First posted 2020-04-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): ePRO intervention + PRAVASTATINE treatment
  Interventions: Other: e-PRO Intervention; Drug: Pravastatin
- CONTROL GROUP (Other): PRAVASTATINE treatment ( without ePRO)
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Other: e-PRO Intervention — Statements of symptoms and patients' health status (PROs) will be collected via a web interface, including access and use in patients with burden symptoms.
  The platform will include four items concerning 7 side effects of fibrosis of grade > 2 in breast cancer. Patients will be encouraged to evaluate on a 5-point Likert scale the frequency, the intensity and the repercussions on the daily life of some symptoms during the last 7 days, in particular on:
  * general pain
  * anxiety
  * sadness
  * texture of the treated breast
  * Patients will also be invited to express themselves on the severity of two other symptoms of their choice, to their worst degree, by listing and rating them on a 5-point scale ranging from "None" to "Very severe" Finally, the aesthetic impact will be evaluated by patients on a visual analogue scale (VAS) of 0 to 100mm
  Other Names: Electronic-Patient Reported Outcomes
  Arms: EXPERIMENTAL GROUP
Drug: Pravastatin — All patients will take Pravastatin 40 mg per day (From Day 0 to Month 12).

SUMMARY:
Conserving surgery followed by adjuvant radiotherapy is currently the therapeutic standard for patient with Breast Cancer. Symptoms are common among patients receiving this treatment. Ten percent of them will develop severe and chronic radio-induced toxicities, such as breast radio-induced-fibrosis impairing their quality of life (QoL). Yet, paying attention to symptom improves the empowerment and psychological adjustment to the disease. Web-based systems that can provide electronic-Patient reported Outcomes (e-PRO) have been shown to prompt clinicians to intensify symptom management, to improve symptom control, and to enhance patient-clinician communication patient satisfaction, as well as well-being.Benefits of systems to elicit e-PRO improve reliable measure of health-related quality of life (QoL) remains discussed.

To date, there are few specific treatments for these severe radio-induced fibrosis except the antifibrotic combinaison Pentoxifylline/Vitamin E with inconsistent result.

Since 2000, we and others have developed a mechanistic approach modulating the severity of RIF by targeting the Rho/ROCK/CTGF pathway, especially by inhibiting Rho activation by pravastatin. Our preclinical data, then followed by the Phase II PRAVACUR-01 trial, concluded that the use of pravastatin has an anti-fibrotic action on different experimental models and reduces the severity of the grade of fibrosis in 50% of patients.

Patients can now benefit from this new anti-fibrotic agent.

Taken as a whole, these data encourage combining both drug (pravastatin) and non-pharmacological intervention , in particular e-PRO, in the RIF management.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients treated by conserving surgery followed by adjuvant RT
2. Over 18 years old
3. At least, grade 2 breast RIF
4. Treatment planning data of breast cancer radiotherapy must be available
5. The following laboratory values obtained ≤ 15 days prior to randomization:

   Serum creatinine ≤ 130 µmol/l; ASAT and ALAT≤ 2N; total bilirubin ≤ 1.5N; CK levels < 3 x ULN, only for the women ≥ 70 years
6. Negative pregnancy test (β-HCG dosage) in women of childbearing potential (women not of reproductive potential are female patients who are postmenopausal or permanently sterilized: e.g., tubal occlusion, hysterectomy, bilateral salpingectomy).
7. Patient without contraindication to treatment with pravastatin
8. Signed and dated written consent
9. Patient must be affiliated to a French Social Security System

Exclusion Criteria:

1. Any breast cancer recurrences
2. Current treatment by : statin, fibrate, ciclosporin, systemic fusidic acid, long-term treatment by corticoids
3. History of muscular dystrophy diseases or chronic and/or hereditary muscular diseases
4. Untreated hypothyroidism
5. Serum creatinine > 130 µmol/l; ASAT and ALAT > 2N; total bilirubin > 1.5N
6. CK levels > 3 x ULN in women over 70 years
7. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody
8. Pregnant or breastfeeding women
9. Women of childbearing potential who are unwilling to employ adequate contraception, from the beginning of the study to 4 weeks after last treatment dose
10. Known hypersensitivity to pravastatin, or any constituent of the product.
11. Patient with alcohol misuse.
12. Patients treated with systemic investigational drugs within the past 30 days
13. Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
evaluate the benefit on breast-related quality of life of systematic e-PROs | From randomization to 12 months
  The BRQoL improvement rate at 12 months, compared with baseline, defined as:
  * an improvement of 5 points (or more) of the score assessed by the functional scale "body image" of the QLQ-BR23 (summary score including the items # 39-42), or
  * a reduction of 5 points (or more) of the score on the symptom scale "breast symptoms" assessed by the QLQ-BR23 (summary score including the items # 51- 53).

SECONDARY OUTCOMES:
evaluate the patients'HRQoL | at baseline;12,24, 36, 48 and 60 months
  defined by the Health-related quality of life assessed by the EORTC QLQ-C30 and its module BR23
estimate the use of antidepressants | From randomization to 12 months
  defined by the rate and dose of used antidepressants
estimate the use of analgesics | From randomization to 12 months
  defined by the rate and dose of used analgesics
estimate the use of anxiolytics | From randomization to 12 months
  defined by the rate and dose of used anxiolytics
Assess the levels of psychological distress | at baseline; at 12, 24, 36, 48 and 60 months
  assessed by (HADS) Scale : score {min :0 (no Distress) --- max :21 ( Hight Distress) }
monitor the e-PROs alerts in the experimental group | From randomization to 12 months
  Timing of the e-PROs alerts and the care management (phone call or planning of a consultation, treatment initiation)
characterise the evaluation of the side effects linked to RIF in the experimental group | From randomization to 12 months
  Evolution of the 7 different e-PROs scores across time (general pain { 0 (no pain)- 4 (high pain)}, anxiety{ 0 (no anxiety)- 4 (high anxiety)}, sadness { 0 (no sad)- 4 (high sad)}, texture of the treated breast{ 0 (no sweeling)- 4 (high sweeling)}, two other symptoms assessed by the PRO-CTCAE scales { 0 (none)- 4 (severe)}, and scores of aesthetic impact assesses by a Visual Analog Scale{ 0 (no impact)- 100 (max impact)}
characterise the modifications of the patients' management in the experimental group | From randomization to 12 months
  Number of hospital emergency visits or hospitalizations
evaluate the anti-fibrotic efficacy of pravastatin | From randomization to 12 months
  Number of supplementary consultations
evaluate the pravastatin safety | From randomization to 12 months
  Regression rate of at least 1 grade of fibrosis (follow-up of fibrosis grade evolution since inclusion)
estimate the relapse-free survival | Until study completion: 5 years
  Relapse-free survival defined as the time from the date of randomization to the date of the first observed oncological event such as local, ipsilateral, regional or metastatic recurrence or death for any cause

CONTACTS AND LOCATIONS:
Locations (1):
- ICM Val d'Aurelle, Montpellier, France